CLINICAL TRIAL: NCT01067287
Title: Blockade of PD-1 in Conjunction With the Dendritic Cell/Myeloma Vaccines Following Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Rambam Health Care Campus (Other); Gateway for Cancer Research (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Avigan, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-061
Record Dates: First submitted 2009-07-29; First posted 2010-02-11 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: dendritic cell fusion vaccine; CT-011; autologous stem cell transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Monoclonal antibody CT-011 will be given 1-3 months following autologous transplant. 3 doses will be given at 6 week intervals.
  Interventions: Drug: CT-011
- Group 2 (Active Comparator): Vaccination with DC/myeloma fusion cells will be given 1-3 months following autologous transplant. Vaccination will be given at 6 weeks intervals. The monoclonal antibody CT-011 will be given 1 week following each vaccination. 3 doses of CT-011 will be given at 6 week intervals.
  Interventions: Drug: CT-011; Biological: Dendritic Cell Fusion Vaccine

INTERVENTIONS:
Drug: CT-011 — Infusions starting one to three months following autologous transplant at 6 week intervals for a total of 3 doses
Biological: Dendritic Cell Fusion Vaccine — One week following each infusion of CT-011
  Arms: Group 2

SUMMARY:
The purpose of this research study is to determine the safety of CT-011 alone, as well as the combination of the Dendritic cell fusion vaccine and CT-011, after autologous stem cell transplantation (ASCT). We are also trying to find out what effect the combination has on the disease, including if it is more successful in preventing or delaying the disease from coming back, compared to treatment with autologous transplantation alone. ASCT is a standard therapy for multiple myeloma that is often successful in significantly decreasing the amount of cancer in the body. CT-011 is an investigational monoclonal antibody. Monoclonal antibodies are a type of drug given by infusion into a vein and are known to target specific cells (in this case, cells in the immune system). The dendritic cell fusion vaccine is an investigational agent that tries to help the immune system to recognize and fight against cancer cells. Unlike a standard vaccine that is used to prevent infections, cancer vaccines are being studied to see if they can fight cancers that are already in the body.

DETAILED DESCRIPTION:
* There are two groups in this study: Group 1: All participants in this study group will receive infusions of CT-011 starting one to three months following autologous transplant. Participants in this group will receive a total of 3 doses of CT-011 at 6 week intervals. Group 2: All participants in this group will receive infusions of CT-011 starting one to three months following autologous transplant. Participants in this group will receive a total of 3 doses of CT-011 at 6 week intervals. In addition, they will receive a vaccination of the Dendritic Cell Fusion Vaccine one week following each infusion of CT-011.
* All participants (Group 1 and Group 2) will receive the following procedures: 1) Initial therapy for multiple myeloma: All participants will receive standard therapy to reduce the number of multiple myeloma cells in the body. 2) Prior to stem cell mobilization participants will undergo a physical exam, medical history, and blood tests to measure blood counts, liver and kidney function, multiple myeloma protein level, and research testing to measure the immune response against the multiple myeloma cells. A small amount of bone marrow will be removed from the participants hip. Participants will also undergo a skin test called "delayed-type hypersensitivity (DTH). 3) Prior to the autologous stem cell transplant, we will harvest stem cells from the participants blood and store then for the future transplant through a process called leukapheresis. 4) Within a few weeks of successful stem cell collection, participants will be admitted to the hospital for high dose chemotherapy with autologous stem cell transplantation (ASCT). 5) Approximately 1-3 months following ASCT, participants will undergo additional tests to assess their eligibility to proceed with treatment with CT-011 alone (group 1) or the combination of CT-011 and vaccination (group 2).
* If the post-transplant eligibility results meet the study requirements participants will receive 3 infusions of CT-011 at 6 week intervals. Prior to each infusion of CT-011, participants will undergo the following procedures: blood tests, urine sample, physical exam and EKG. Participants will be seen weekly to review any side effects, what medications they are taking, and will have a blood test an physical exam.
* For Group 2 participants only: Prior to autologous transplant, Group 2 participants will undergo several procedures to make the Dendritic Cell Fusion Vaccine. 1) Dendritic Cell Collection via leukapheresis 2) Tumor cell collection from the participants bone marrow. One week after receiving the CT-011 infusion, Group 2 participants will receive the study vaccine for a total of 3 vaccines.
* After the final treatment both Group 1 and Group 2 participants will receive a tumor DTH injection and DTH to Candida into the skin. At one, three and six months following the last study treatment participants will have blood tests, urine test, bone marrow aspirate/biopsy and a skeletal survey. At two, four and five months, participants will have a blood test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma who are potential candidates for high doses chemotherapy with stem cell rescue
* Patients must not have active of history of autoimmune disorders/conditions including Type I diabetes, Type II diabetes, vitiligo or stable hypothyroidism will not be considered exclusion criteria
* Patients with measurable disease as defined by a history of an elevated M component in plasma, urine, or free kappa/lambda light chains in the serum
* 18 years of age or older
* ECOG Performance Status of 0-1 with a greater than nine week life expectancy
* >20% bone marrow involvement in plasmacytoma amenable to resection under local anesthesia
* Negative pregnancy test and adequate contraception method(s)
* DLCO (adjusted) > 50%
* Cardiac Ejection Fraction > 45%
* Laboratory results as defined in protocol

Exclusion Criteria:

* History of clinically significant venous thromboembolism
* Clinically significant autoimmune disease
* HIV positive
* Serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, ischemic coronary disease or congestive heart failure
* Pregnant or lactating women
* History of allogeneic bone marrow/stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2010-03; Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
First Stage: To explore immunological response to CT-011 in the post transplant period. | 3 years
Second Stage: To determine if cellular immunity is induced by treatment with monoclonal antibody CT-011 and DC/myeloma fusion cells in conjunction with stem cell transplant. | 3 years

SECONDARY OUTCOMES:
First Stage: To assess the toxicity associated with treating multiple myeloma patients with CT-011 in the post- autologous transplant setting. | 3 years
Second Stage: To assess the toxicity associated with treating multiple myeloma patients with the combination with DC/myeloma fusion vaccine following autologous transplant. | 3 years
Second Stage: To correlate levels of circulating activated and regulatory T cells with immunologic response | 3 years
Second Stage: To define anti-tumor effects using serum markers, radiological studies, and time to progression. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Rambam Medical Center, Haifa, Israel